CLINICAL TRIAL: NCT03915236
Title: Prospective, Randomized, Open, Controlled, Multicenter Study to Evaluate the Safety and Efficacy of the MON4STRAT Approach for Optimizing Meropenem Therapy in Intubated and Mechanically-Ventilated, Adult Patients With Severe Gram-Negative Lower Respiratory Tract Infection MON4STRAT Study
Brief Title: Approach for Optimizing Meropenem Therapy in Intubated and Mechanically-Ventilated, Adult Patients With Severe Gram-Negative Lower Respiratory Tract Infection
Acronym: MON4STRAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was decided to discontinuate the study due to a very low recruitment.
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MON4STRAT; 2018-000450-21 (EudraCT Number)
Record Dates: First submitted 2019-04-03; First posted 2019-04-16 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2019-04

CONDITIONS: Lower Respiratory Tract Infection
Keywords: MON4STRAT; Treatment Drug Monitoring; Antibiotic Resistance; Beta-Lactams Resistance; Meropenem; Health Care-Asociated Infection
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: MON4STRAT Strategy (Experimental)
  Interventions: Device: MON4STRAT Strategy
- Group 2: Conventional treatment (Active Comparator)
  Interventions: Other: Control group

INTERVENTIONS:
Device: MON4STRAT Strategy — Meropenem infusion guided by daily Therapeutic Drug Monitoring (adjusted in order to reach predetermined PK/PD targets) using MON4STRAT device.
  Arms: Group 1: MON4STRAT Strategy
Other: Control group — Meropenem 1 gram infused every 8 hours over 30 minutes, consistent with standard-of-care treatment and published guidelines. Meropenem doses will be modified according to SmPC recommendations.
  Arms: Group 2: Conventional treatment

SUMMARY:
Antibacterial drugs are facing increasing limitations in terms of effectiveness due to emergence resistance. Improved antibacterial drug monitoring approaches are particularly needed in nosocomial infections occurring in ICU patients, including ventilator-associated pneumonia and ventilator-associated tracheobronchitis, where decreased susceptibility of the etiological organisms is observed worldwide and pharmacokinetic alterations frequently observed.

No routine drug monitoring is available for betalactams at the point of care in a useful time frame (i.e., within a few hours after having collected the blood specimens).

The purpose of this study is to compare MON4STRAT approach for reaching and maintaining a meropenem pre-determined PK-PD target when compared to conventional meropenem dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females, 18 years of age or older
2. Currently intubated and mechanically-ventilated subjects in the ICU
3. Suspicion of lower respiratory tract infection
4. Presence of Gram-negative organism(s) by Gram stain OR by culture of pre-therapy respiratory specimen (eg, endotracheal aspirate [ETA], bronchoalveolar lavage [BAL], or mini-BAL) OR previous colonization 48 h before screening.
5. Initial empiric antimicrobial meropenem regimen
6. At least two risk factors for multidrug-resistant organisms
7. Provision of written informed consent by the subject or a family member or a close relative or waiver of consent.

Exclusion Criteria:

1. Subjects who have received antibiotic therapy for Gram-negative LRT infection for ≥ 36 hours at the time of randomization
2. Subjects with known or suspected type 1 hypersensitivity to beta-lactam and/or cephalosporin
3. Subjects taking valproic acid for a seizure disorder
4. Subjects who have had a left hemisphere stroke within five days and there is an increased risk of fatal brain oedema
5. Subjects who have cystic fibrosis, human immunodeficiency virus (HIV) infection with CD4 count <100 cell/mm3 or invasive fungal infection of the lung
6. Neutropenia (ANC < 103 neutrophils/mm3)
7. Bone marrow transplant.
8. Subjects who have been on mechanical ventilation for >28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
To document the superiority of the MON4STRAT approach for reaching and maintaining a meropenem pre-determined PK-PD target when compared to conventional therapies. | During meropenem treatment: Day1 to Day 7
  The proportion of time from day 1 after randomization to end of therapy (EOT) in which the free meropenem trough concentration in serum was maintained above 8 mg/L or above 4 x MIC if antibiotic MIC > 2 and ≤ 8 mg/L, without exceeding 140 mg/L at peak level, as determined by a method of reference (HPLC).

SECONDARY OUTCOMES:
Clinical and microbiological response rates | Test of cure (TOC) visit (7 to 10 days after last study drug infusion)
Time to LRT bacterial eradication, as assessed by follow-up cultures of ETA | Days 3, 5, 7 of treatment and at the end of treatment (EOT) visit
All-cause mortality | Day 14 and day 28
ICU and hospital length of stay | Up to day 28
Number of mechanical ventilation-free days, defined as the number of days of unassisted breathing | Up to day 28

CONTACTS AND LOCATIONS:
Locations (3):
- Université Libre de Bruxelles, Brussels, Belgium
- Pitié Salpêtrière Hospital, Paris, France
- Hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No